CLINICAL TRIAL: NCT03004794
Title: Characteristics and Predictors of Progression of an Egyptian Multiple Sclerosis Cohort
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hatem Samir Shehata, Professor of Neurology, Cairo University
Other Study IDs: RC4
Record Dates: First submitted 2016-12-15; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Other: medical records review

SUMMARY:
Initial recruitment: 1717, 136 (7.92%) were excluded due to missing data that could not be obtained. The diagnosis of multiple sclerosis (MS) was revised according to the 2010 revision of the McDonald criteria.

Patients analyses: 1581 Every patient was registered by his/her 14-digit unique identity numbers, (which is mandatory in Egypt since 1999) to make sure that every registered patient in different centers were counted only once.

DETAILED DESCRIPTION:
Patients' records review procedure and sampling strategies. The medical records, administrative data, laboratory and diagnostic tests reports were screened by 3 authors (HS, NS, AE) and these data were extracted in a standard electronic form according to Kasr Alaini Multiple Sclerosis Unit (KAMSU) registry.

An assigned coordinator from each center was requested to facilitate data collection from site-specific records. In cases of incomplete documentation or unclear information, verification was done by on-site data coordinator either by phone contact or face-to-face interview with the patients, whether during the routine follow up or in an unscheduled visit.

Several measures were taken to ensure the confidentiality of the collected information. No patient names were included in the database presented by site coordinator, and the study staff signed a confidentiality agreement for non-disclosure.

ELIGIBILITY:
Inclusion Criteria:

* All patients with suspecting multiple sclerosis attending 4 tertiary referral centers in Egypt

Exclusion Criteria:

* missing data that could not be obtained

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The diagnosis of multiple sclerosis (MS) was revised according to the 2010 revision of the McDonald criteria, and patients were classified according to the course of the disease into relapsing remitting multiple sclerosis (RRMS), secondary progressive multiple sclerosis (SPMS) and primary-progressive multiple sclerosis (PPMS). Patients with first demyelinating event, before 2010, were re-assessed by on-site coordinators to label them clinically isolated syndrome (CIS), whenever applicable, according to McDonalds 2010, and neuromyelitis optica (NMO) cases diagnosis was verified according to the 2015 diagnostic criteria. Those with typical brain Magnetic Resonant Imaging (MRI) MS like lesions without related clinical manifestations were diagnosed as radiologically isolated syndrome (RIS).
Sampling Method: Probability Sample
Enrollment: 1581 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Evoked Potentials (measure latency in m.sec) | 13 months (through study completion)
  Number of patients with delayed latency of Evoked Potentials
Cerebrospinal Fluid (CSF): measure IgG index and Oligoclonal bands (OCB) | 13 months (through study completion)
  Number of patients with elevated IgG index and OCB